CLINICAL TRIAL: NCT01417741
Title: Is Intra-operative Acupuncture at P6 Plus IV Antiemetics More Effective Than IV Antiemetic Therapy Alone in Preventing Postoperative Vomiting in Pediatric Patients Following Tonsillectomy With or Without Adenoidectomy?
Brief Title: Acupuncture and Nausea/Vomiting in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Angela Kendrick, associate professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: APOM-7605
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Vomiting and Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy Only (No Intervention): Patients will not receive acupuncture. Standard anti-emetic therapy will be given.
- Acupuncture Plus Standard Therapy (Experimental): Bilateral P6 acupuncture applied after anesthesia induction and removed at the termination of the surgery. Patients will also receive standard anti-emetic therapy.
  Interventions: Device: Acupuncture Needle

INTERVENTIONS:
Device: Acupuncture Needle — A small 1.8 mm needle to be placed in the P6 acupuncture point on the wrist
  Other Names: Seirin Pyonex
  Arms: Acupuncture Plus Standard Therapy

SUMMARY:
The purpose of this study is to investigate the effects of intraoperative P6 acupuncture plus standard therapy on postoperative nausea and vomiting in pediatric patients undergoing tonsillectomy with or without adenoidectomy. 200 children will be randomly assigned to either the treatment or the control group.

1. Treatment Group: Standard anti-emetic therapy plus bilateral P6 acupuncture after the induction of anesthesia
2. Control Group: Standard anti-emetic therapy only

This study will monitor nausea, retching, and vomiting events both directly after the surgery as well as the next day via a follow-up phone call to the parents of the study participant.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 to 3 physical status
* Undergoing Tonsillectomy and/or adenoidectomy
* Consent obtained from Parent/Guardian

Exclusion Criteria:

* Taking preoperative steroids, including inhalers
* Taking baseline anti-emetics
* History of motion sickness
* BMI > 35 (morbid obesity)
* Severe OSA (Apnea/hypopnea Index > 10)
* Have genetic abnormalities

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Kendrick, MD, Principal Investigator — Oregon Health and Science University; Christine Martin, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Sciences University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin CS, Deverman SE, Norvell DC, Cusick JC, Kendrick A, Koh J. Randomized trial of acupuncture with antiemetics for reducing postoperative nausea in children. Acta Anaesthesiol Scand. 2019 Mar;63(3):292-297. doi: 10.1111/aas.13288. Epub 2018 Nov 6. PMID 30397904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: randomization of three patients unrecorded, so 161 properly randomized patients were entered in study
Groups:
- Standard Therapy Only: Patients will not receive acupuncture. Standard anti-emetic therapy will be given.
  Standard anti -emetic therapy at our institution for children having a T and A consists of Ondansetron 0.15 mg/kg and dexamethasone 0.25mg/kg up to 10 mg.
Period: Overall Study
Arm/Group | Standard Therapy Only | Acupuncture Plus Standard Therapy
Started | 75 | 86
Completed (Of the children who received the standard therapy, only 69 recived the post op day one phone call.) | 75 | 86 (only 73 received the post op day phone phone call)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Therapy Only: Patients will not receive acupuncture. Standard anti-emetic therapy will be given.
  Children ages 3-9 undergoing tonsillectomy with or without adenoidectomy were the population studied in both arms.
- Total: Total of all reporting groups
Arm/Group | Standard Therapy Only | Acupuncture Plus Standard Therapy | Total
Number analyzed (Participants) | 75 | 86 | 161
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 5.5 (1.8) | 5.2 (1.9) | 5.3 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 45 | 78
  Male | 42 | 41 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Study took place at DCH ( Children's hospital ) in Portland OR
  participants
    United States | 75 | 86 | 161

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Nausea and Vomiting
Description: Post operative Nausea and vomiting in phase 1 and 11 recovery (Measured as a percentage of participants who experienced this outcome) Post op Nausea and vomiting on post op day one ( measured as a percentage of participants who experienced this outcome) as reported on a telephone survey
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Groups:
- Standard Therapy Only: Patients will not receive acupuncture. Standard anti-emetic therapy will be given.
  In phase i and 11 recovery units 26 patients ( 34.7 %) of 75 patients in this arm experienced Nausea and or vomiting.
  on POD 1; 37 patients or 54% experienced nausea or vomiting
- Acupuncture Plus Standard Therapy: Bilateral P6 acupuncture applied after anesthesia induction and removed at the termination of the surgery. Patients will also receive standard anti-emetic therapy.
  Acupuncture Needle: A small 1.8 mm needle to be placed in the P6 acupuncture point on the wrist
  In phase 1 and 11 recovery units: 6 patients ( 7%) of 86 experienced nausea or vomiting On POD one: 31 or 43% experienced PONV
Arm/Group | Standard Therapy Only | Acupuncture Plus Standard Therapy
Number analyzed (Participants) | 75 | 86
Participants
  Immediate Post Op | 26 | 6
  Post Op Day 1 | 37 | 31

ADVERSE EVENTS:
Time Frame: Post-operative day (POD) 0 and day 1
Groups:
- Standard Therapy Only ( AE Group): Patients will not receive acupuncture. Standard anti-emetic therapy will be given.
Arm/Group | Standard Therapy Only ( AE Group) | Acupuncture Plus Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/86
Other Adverse Events (participants affected / at risk) | 0/75 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No